CLINICAL TRIAL: NCT04313933
Title: Plasma Citrulline in Preterm With NEC
Acronym: NEC
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Mostafa, Principal Investigator, Ain Shams University
Other Study IDs: FMASU M S 419/2019
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-02

CONDITIONS: NEC; Citrulline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of study

DETAILED DESCRIPTION:
Introduction

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates < 35 weeks Preterm neonates< 2kg Preterm neonates diagnosed with necrotizing enterocolitis

Exclusion Criteria:

* renal dysfunction Inborn error of metabolism Congenital malformation

Ages: 1 Day to 30 Days | Sex: All
Age Groups: Child
Study Population: Preterm neonates admitted to NICU at Ain Shams Unversity Hospitals
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
plasma citrulline as a marker of Necrotizing enterocolitis diagnosis | 1 Year
  Compare plasma citrulline in NEC and comparing it with properly matched healthy neonates

SECONDARY OUTCOMES:
Citrulline as a marker of intestinal recovery | 1 year
  Follow up plasma citrulline level after initiation of feeding

CONTACTS AND LOCATIONS:
Overall Officials: Amira Mostafa, Study Director — Ain Shams University
Locations (1):
- AinShams University, Cairo, Egypt